CLINICAL TRIAL: NCT05430022
Title: Adapted Cognitive Behavioral Therapy for Depression in Autistic Youth: A Pilot Trial
Brief Title: Group Depression Treatment for Autistic Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Schwartzman, PhD, Assistant Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201725
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder; Depression; Suicidal Ideation; Self Esteem
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Pilot, nonrandomized trial of a behavioral intervention for autistic adolescents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism-adapted Group Cognitive Behavioral Therapy (Child Ratings) (Experimental): Autistic adolescents (11-17 years old; middle and high school) with depression will participate in a 12-week group intervention, autism-adapted Cognitive Behavioral Therapy, to increase perception and understanding of self and to decrease the severity of depressive symptoms.
  Interventions: Behavioral: Autism-adapted Group Cognitive Behavioral Therapy
- Autism-adapted Group Cognitive Behavioral Therapy (Parent Ratings) (Experimental): One parent of each autistic adolescent (11-17 years old; middle and high school) with depression will provide ratings of their child as their child participates in a 12-week group intervention, autism-adapted Cognitive Behavioral Therapy, to decrease the severity of depressive symptoms. Parents will not participate in therapy sessions.
  Interventions: Behavioral: Autism-adapted Group Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Autism-adapted Group Cognitive Behavioral Therapy — The autism-adapted Group Cognitive Behavioral Therapy (CBT) was designed by the PI and research team in collaboration with autistic stakeholders (i.e., adults, parents, researchers). It is a 12-week group intervention (90 min) delivered on a weekly basis in an outpatient psychiatry clinic by licensed clinical psychologists and psychology trainees. Each group is comprised of 8-9 autistic adolescents (11-17 years old; middle and high school) with depression. The intervention targets adolescents' perception and understanding of self, including autistic identity, through a series of cognitive-behavioral approaches including psychoeducation, emotion regulation, cognitive distortions, cognitive restructuring, behavioral rehearsals, and weekly homework assignments.

SUMMARY:
Higher rates of depression are reported by autistic adolescents as compared to their non-autistic peers, which is problematic given adverse outcomes (e.g., negative self-esteem, lower academic performance) that are associated with depression. Despite the alarming rates of depression in autistic youth and associated safety concerns, few treatments have been developed. In this study, we investigate the feasibility, acceptability, and preliminary efficacy of an autism-adapted group cognitive-behavioral treatment for autistic adolescents (11-17 years old; middle and high school) in a pilot, nonrandomized trial. Specifically, we aim to increase adolescents' perception and understanding of self, including autistic identity, in order to treat depression. Intervention design and implementation were guided by autistic self-advocates and parents.

DETAILED DESCRIPTION:
Higher rates of depression and suicidal thoughts are reported by autistic adolescents as compared to their non-autistic peers, which is problematic given adverse outcomes (e.g., negative self-esteem, lower academic performance) that are associated with depression. Despite the alarming rates of depression in autistic youth, few interventions have been developed or tested to reduce depression in this at-risk population. An evidence-based intervention for depression in non-autistic adolescents is Cognitive Behavioral Therapy (CBT), which CBT has strong research support for treating depression in non-autistic adolescents according to the American Psychological Association (APA). Autism-adapted CBT programs for anxiety and OCD have outperformed standard CBT approaches for autistic youth; however, autism-adapted CBT programs for depression in autistic adolescents have not been developed with stakeholders nor tested in a clinical setting. To address this gap, an adapted CBT group intervention for autistic adolescents (11-17 years old; middle and high school) with depression was designed in collaboration with autistic stakeholders.

In the present study, the feasibility, acceptability, and preliminary efficacy of this 12-week group intervention in improving perception and understanding of self and depressive symptoms will be examined in a pilot, nonrandomized trial with pretest-posttest design. Groups will occur in the Outpatient Clinic of the Department of Psychiatry and Behavioral Sciences at the Vanderbilt University Medical Center (VUMC), and study measures will be administered to adolescents and their parents at four timepoints: baseline (week 0), midpoint (week 6), post (week 12), and follow-up (week 24). Study measures include parent- and self-report measures of adolescent well-being (e.g., perception of self, quality of life, etc.) and clinical interviews of psychiatric symptoms (e.g., depressive symptoms, suicidal thoughts). The significance and size of intervention effects on emotional and behavioral outcomes will be measured using one-way ANOVAs and linear mixed models. If predicted results occur, it will provide information on the feasibility and acceptability of this group intervention, with preliminary empirical support for its efficacy in improving perception and understanding of self and reducing the severity of depressive symptoms in autistic adolescents.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* 11 to 17 years of age (middle or high school)
* Diagnosis of Autism Spectrum Disorder
* Average to above-average intellectual functioning
* Willing to attend study visits and participate in weekly group intervention

Adolescent Exclusion Criteria:

* No diagnosis of Autism Spectrum Disorder
* Comorbid intellectual impairment (FSIQ < 70), as the study protocol and assessments are not designed, and thus not appropriate, for this population.
* Severe medical conditions (e.g., uncontrolled seizures) and/or genetic disorders (e.g., Fragile X syndrome).
* Unwilling to attend study visits or weekly group intervention sessions.
* Significant aggression to self/others
* Significant active suicidal thoughts with intent/plan requiring higher-level care

Parent Inclusion Criteria:

* At least 18 years of age and a parent or legal guardian of the adolescent participant with ASD.
* Able to provide current and historical observations of the functioning of the participant with ASD based on self report from parent. Similarly, parent must live in close proximity to and have frequent contact with the participant with ASD.
* Willing to complete questionnaires about their own functioning and that of their child with ASD.

Parent Exclusion Criteria:

-Parents of adolescents with ASD who do not have frequent contact with the participant with ASD and/or unable to provide current and historical observations of the functioning of the participant with ASD.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Schwartzman, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Autism-adapted Group Cognitive Behavioral Therapy (Child Ratings): Autistic adolescents (11-17 years old; middle and high school) with depression will participate in a 12-week group intervention, autism-adapted Cognitive Behavioral Therapy, to decrease the severity of depressive symptoms.
  Autism-adapted Group Cognitive Behavioral Therapy: The autism-adapted Group Cognitive Behavioral Therapy (CBT) was designed by the PI and research team in collaboration with autistic community members (i.e., adults, parents, researchers). It is a 12-week group intervention (90 min) delivered on a weekly basis in an outpatient psychiatry clinic by licensed clinical psychologists and psychology trainees. Each group is comprised of 8-9 autistic adolescents (11-17 years old; middle and high school) with depression. The intervention targets adolescents' perception and understanding of self, including autistic identity, through a series of cognitive-behavioral approaches including psychoeducation, emotion regulation, cognitive distortions, cognitive restructuring, behavioral rehearsals, and weekly homework assignments.
- Autism-adapted Group Cognitive Behavioral Therapy (Parent Ratings): One parent of each autistic adolescent (11-17 years old; middle and high school) with depression will provide ratings of their child as their child participates in a 12-week group intervention, autism-adapted Cognitive Behavioral Therapy, to decrease the severity of depressive symptoms. Parents did not participate in therapy sessions.
  Autism-adapted Group Cognitive Behavioral Therapy: The autism-adapted Group Cognitive Behavioral Therapy (CBT) was designed by the PI and research team in collaboration with autistic community members (i.e., adults, parents, researchers). It is a 12-week group intervention (90 min) delivered on a weekly basis in an outpatient psychiatry clinic by licensed clinical psychologists and psychology trainees. Each group is comprised of 8-9 autistic adolescents (11-17 years old; middle and high school) with depression. The intervention targets adolescents' perception and understanding of self, including autistic identity, through a series of cognitive-behavioral approaches including psychoeducation, emotion regulation, cognitive distortions, cognitive restructuring, behavioral rehearsals, and weekly homework assignments.
Period: Overall Study
Arm/Group | Autism-adapted Group Cognitive Behavioral Therapy (Child Ratings) | Autism-adapted Group Cognitive Behavioral Therapy (Parent Ratings)
Started | 24 | 24
Completed | 20 | 20
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: 24 child and parent dyads
Groups:
- Total: Total of all reporting groups
Arm/Group | Autism-adapted Group Cognitive Behavioral Therapy (Child Ratings) | Autism-adapted Group Cognitive Behavioral Therapy (Parent Ratings) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 0 | 24
  Between 18 and 65 years | 0 | 24 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.79 (1.96) | 48.32 (5.78) | 31.06 (3.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 19 | 28
  Male | 15 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48
Social Responsiveness Scale, Second Edition [Mean (Standard Deviation); unit: T-score] — The SRS-2 measures an individual's degree of social impairment and restricted, repetitive behaviors and/or interests in the past six months. Raw scores are converted to T-scores with a mean of 50 and a standard deviation of 10, with higher scores indicating more impairment. T-scores between 60-64 indicate "mild" social impairment and restricted, repetitive behaviors and/or interests, T-scores between 65-75 indicate "moderate" impairment, and T-scores at/above 76 indicate "severe" impairment on the SRS-2. Data were not collected for the parent population. Population: data were not collected for the parent population
  T-score
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 75.64 (9.1) |  | 75.64 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Adolescent Depressive Symptoms, Self-report
Description: Self-reported severity of depressive symptoms by autistic adolescents on the Revised Children's Anxiety and Depression Scale (RCADS). The RCADS is a 47-item scale with each item scored from 0-3, with a total possible raw score of 0-141, with higher scores indicating higher internalizing symptoms. The depression subscale of the RCADS is comprised of 10 items. Raw scores are converted to grade-based standardized T-scores (mean of 50, standard deviation of 10), and T-scores greater than 59 indicate clinically-significant symptoms. The RCADS has been validated for use with autistic youth.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Autism-adapted Group Cognitive Behavioral Therapy: Autistic adolescents (11-17 years old; middle and high school) with depression will participate in a 12-week group intervention, autism-adapted Cognitive Behavioral Therapy, to decrease the severity of depressive symptoms.
  Autism-adapted Group Cognitive Behavioral Therapy: The autism-adapted Group Cognitive Behavioral Therapy (CBT) was designed by the PI and research team in collaboration with autistic community members (i.e., adults, parents, researchers). It is a 12-week group intervention (90 min) delivered on a weekly basis in an outpatient psychiatry clinic by licensed clinical psychologists and psychology trainees. Each group is comprised of 8-9 autistic adolescents (11-17 years old; middle and high school) with depression. The intervention targets adolescents' perception and understanding of self, including autistic identity, through a series of cognitive-behavioral approaches including psychoeducation, emotion regulation, cognitive distortions, cognitive restructuring, behavioral rehearsals, and weekly homework assignments.
Arm/Group | Autism-adapted Group Cognitive Behavioral Therapy
Number analyzed (Participants) | 20
T-score | 8.14 (2.1)

2. Primary Outcome: Change in Severity of Adolescent Depressive Symptoms, Parent-report
Description: Parent-reported severity of adolescent depressive symptoms on the Revised Children's Anxiety and Depression Scale (RCADS). The RCADS is a 47-item scale with each item scored from 0-3, with a total possible raw score of 0-141, with higher scores indicating higher internalizing symptoms in adolescents. The depression subscale of the RCADS is comprised of 10 items. Raw scores are converted to grade-based standardized T-scores (mean of 50, standard deviation of 10), and T-scores greater than 59 indicate clinically-significant symptoms. The RCADS has been validated for use with autistic youth.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Autism-adapted Group Cognitive Behavioral Therapy
Number analyzed (Participants) | 20
T-score | 3.42 (2.2)

ADVERSE EVENTS:
Time Frame: Baseline to 6-months after baseline visit at end of study participation.
Description: Systematic assessment of adolescent suicidal thoughts and/or behaviors and severity of depressive symptoms, per self- and parent-report. Assessments collected at four timepoints between the baseline study visit and 6-month follow-up study visit (i.e., end of study participation).
Arm/Group | Autism-adapted Group Cognitive Behavioral Therapy (Child Ratings) | Autism-adapted Group Cognitive Behavioral Therapy (Parent Ratings)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT05430022/Prot_001.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT05430022/SAP_002.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT05430022/ICF_000.pdf